CLINICAL TRIAL: NCT03147963
Title: A Randomized, Controlled Clinical Trial Comparing the Efficacy and Safety of a Single Agent Docetaxel 2-weeks Regimen in the Treatment of HER2 Negative Metastatic Breast Cancer to a 3-weeks Regimen
Brief Title: Docetaxel 2-weeks Regimen in the Treatment of HER2 Negative Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Huang Ping, attending doctor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZCHBC0011
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: therapy; breast cancer; docetaxel; metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: patients was divided 1:1 into docetaxel 2-weeks regimen group and docetaxel 3-weeks regimen group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Docetaxel 2-Weeks regimen group (Experimental): Docetaxel injection 50mg/m2,iv,d1,every 2 weeks
  Interventions: Drug: Docetaxel
- Docetaxel 3-Weeks regimen group (Active Comparator): Docetaxel injection 75mg/m2,iv,d1,every 3 weeks
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be given until progression or patient intolerance

SUMMARY:
A Randomized, Controlled Clinical Trial Comparing the Efficacy and Safety of a Single Agent Docetaxel 2-Weeks Regimen in the Treatment of HER2 Negative Metastatic Breast Cancer to a 3-Weeks Regimen

DETAILED DESCRIPTION:
Docetaxel 2-Weeks Regimen:Docetaxel 50mg/m2 Docetaxel 3-Weeks Regimen:Docetaxel 75mg/m2

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* The age is Above 18 years of age, <70 years old
* The diagnosis of breast cancer was confirmed by cytological examination or pathological examination. HER2-negative
* Clinical stage was metastatic breast cancer or locally advanced breast cancer.
* Must have at least one measurable lesion, according to RECISTv1.1.
* Eastern Cooperative Oncology Group performance status (ECOG PS)=0~2
* Docetaxel or paclitaxel can been used in initial treatment or in the past for locally advanced, recurrent or metastatic lesions,if used must been proved effective, and recent progress over 6 months.
* The basic function of normal bone marrow
* Functions of liver and kidney is normal
* Expectation of life is more than 3 months
* Agreed to take contraceptive measures during treatment

Exclusion Criteria:

* The patient had a history of allergy to taxanes or their components.
* Recent progress of taxanes in 6 months.
* In the elution period of other chemotherapy regimens.
* Severe coagulopathy.
* HER2 positive breast cancer
* Previous toxicity was not recovered to 0-1 degrees
* Central nervous system metastasis had not Controlled yet
* Pregnancy or lactation
* There are uncontrolled infection, myocardial infarction, thrombosis, etc.
* There are uncontrolled chronic diseases such as diabetes, hypertension, peptic ulcer, chronic hepatitis, mental disease;
* HIV infection
* Patients with other malignant tumor history, except the healed skin basal cell carcinoma and carcinoma of uterine cervix;
* Researchers believe that is not suitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-12-20 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 5 years
  Progression-free survival (PFS) is defined as the time elapsed between enrolling and tumor progression or death from any cause

SECONDARY OUTCOMES:
Overall survival(OS) | From date of enrolling until the date of death from any cause, assessed up to 5 years
  The time elapsed between enrolling and death from any cause
Clinical benefit rate(CBR) | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 5 years
  The response is CR+PR+SD ≥ 24 weeks
Quality of life（QOL） | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first，assessed up to 5 years
  Score change from enrolling to progression disease or death according EORTC QLQ-C30.The EORTC QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients.
Number of participants with Grade 3/4 adverse events | From date of enrolling until the date of 1 month of stop treatment, assessed up to 5 years
  Number of participants with Grade 3/4 adverse events of the two groups was assessed in accordance with the common terminology criteria (NCI CTC AE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojia WANG, MD,PHD, Principal Investigator — Zhejiang Cance Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nabholtz JM, Falkson C, Campos D, Szanto J, Martin M, Chan S, Pienkowski T, Zaluski J, Pinter T, Krzakowski M, Vorobiof D, Leonard R, Kennedy I, Azli N, Murawsky M, Riva A, Pouillart P; TAX 306 Study Group. Docetaxel and doxorubicin compared with doxorubicin and cyclophosphamide as first-line chemotherapy for metastatic breast cancer: results of a randomized, multicenter, phase III trial. J Clin Oncol. 2003 Mar 15;21(6):968-75. doi: 10.1200/JCO.2003.04.040. PMID 12637459